CLINICAL TRIAL: NCT03472079
Title: Does the Urine Concentration of TIMP2*IGFBP7 Can Distinguish Patients Who Will Present Transient or Persistent Acute Kidney Injury During Septic Shock? A Retrospective Analysis. BIOCHECK
Brief Title: TIMP2*IGFBP7 and Transient AKI
Acronym: BIOCHECK
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0013
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Septic Shock
Keywords: Acute kidney injury; Septic shock; TIMP2*IGFBP7
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with septic shock in the intensive care unit have a high risk to develop acute kidney injury (AKI) and AKI is an independent risk factor of mortality. Given the absence of validated pharmacological treatments for limiting the progression of AKI or for accelerating recovery from AKI, early intervention and the restoration of the glomerular filtration rate (GFR) in this context of septic shock might improve the patients' prognosis. One major challenge is to determine whether or not the AKI is reversible (return to normal function KDIGO 0 within 72 hours). In this retrospective study the investigators will analyze all patients admitted for a septic shock in three French ICUs between the 1st january 2014 and 01st January 2017 who developed an AKI (KDIGO ≥1) at admission and who had a determination of the urine concentration of TIMP2*IGFBP7 at admission. The investigators will determine the best threshold of TIMP2*IGFBP7 to distinguish the population of patients who will return to normal kidney function within 72 hours (KDIGO 0).

DETAILED DESCRIPTION:
Background :

Patients with septic shock in the intensive care unit have a high risk to develop acute kidney injury (AKI). AKI is an independent risk factor of mortality. Given the absence of validated pharmacological treatments for limiting the progression of AKI or for accelerating recovery from AKI, early intervention and the restoration of the glomerular filtration rate (GFR) in this context of septic shock might improve the patients' prognosis. One major challenge is therefore how to determine whether or not the AKI is reversible. The best-studied biomarkers (NGAL and KIM 1) have little discriminant power in septic patients because of their poor specificity or unsuitable kinetics for very early diagnosis. The combination of urine assays for tissue inhibitor of metalloproteinase 2 (TIMP2) and insulin-like growth factor binding protein 7 (IGFBP7) has shown good diagnostic performance for the very early detection of the risk of developing AKI in the following 12 hrs. Urine levels of these two markers specifically reflect damage to kidney tubules. Moreover, the levels appear to be strongly correlated with the severity of tubule damage. Thus, one can reasonably hypothesize that measurement of these markers in the very early stages of septic shock might determine the presence and severity of kidney tubule damage. A threshold (yet to be defined) would help to differentiate between (i) transient, non-severe injury and (ii) injury that is already too severe to be reversible.

Purpose : to determine whether or not the urine concentration of TIMP2*IGFBP7 may distinguish patients with high risk of persistent or transient AKI during the early phase of septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Inclusion criteria: septic shock (according to Bone's criteria) within 4 hours following the introduction of catecholamines, AKI defined by KDIGO≥1, social security coverage, measurement of the urine concentration of TIMP2*IGFBP7 within the 4 hours following the introduction of catecholamines, patients admitted for a septic shock between 1st January 2014 and 1st January 2017 in the medical ICU of Amiens university hospital France, medical ICU of Montpellier university hospital France and ICU Melun hospital, France

Exclusion Criteria:

* Need for immediate renal replacement therapy, anuria, chronic renal failure (stage 4 or 5 with GFR<30ml/min), obstructive AKI, pregnancy, cardiac arrest during the same hospitalization, life expectancy<48 hours, Child C Cirrhosis, prior occurrence of AKI during the current hospital stay, kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: univariate comparison between the 2 groups (transient and persistent AKI) using Mann Whithney test or Chi square test. ROC curve analysis to determine the best threshold of TIMP2*IGFBP7 groups to distinguish the 2 groups.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
KDIGO value | return to KDIGO 0 within the first 72 hours following the introduction of catecholamines
  : Transient AKI defined by the return to KDIGO 0 within the first 72 hours following the introduction of catecholamines

SECONDARY OUTCOMES:
need for renal replacement therapy | within the first 72 hours following the introduction of catecholamines
  need for renal replacement therapy within the first 72 hours following the introduction of catecholamines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France